CLINICAL TRIAL: NCT05670938
Title: Follow-up After Surgery for Testicular Cancer: the Prospective, Single Centre FUTURE-testis Implementation Study
Brief Title: Follow-up After Surgery for Testicular Cancer
Acronym: FUTURE-testis
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, D.J. (Dirk) Grünhagen, Principal Investigator, Erasmus Medical Center
Other Study IDs: NL78539.078.21
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Testicular Cancer; Testicular Germ Cell Tumor; Quality of Life
Keywords: Follow-up
MeSH Terms: conditions — Testicular Neoplasms; Testicular Germ Cell Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-seminomatous germ cell tumours, stage I low risk: No lymphadenopathy or metastases on the postoperative scan. Three consecutive blood drawings with normal tumour markers. Patients undergoing lymph node dissection as a second curative operation after an orchiectomy, can also be included in case that the postoperative scan shows no residual disease or metastases.
- Non-seminomatous germ cell tumours, stage I high risk: After completion of one cycle of Bleomycin, etoposide and platinum (BEP). Biochemical remission at completion of chemotherapy, meaning three consecutive blood drawings with normal tumour markers.
  No lymphadenopathy or metastases on the CT scan after completion of chemotherapy.
- Seminomatous germ cell tumours (after chemotherapy) with complete remission.: Biochemical remission at completion of chemotherapy, meaning three consecutive blood drawings with normal tumour markers.
  No lymphadenopathy or metastases on the CT scan after completion of chemotherapy.
- Non-seminomatous germ cell tumours (after chemotherapy) with complete remission.: Biochemical remission at completion of chemotherapy, meaning three consecutive blood drawings with normal tumour markers.
  No lymphadenopathy or metastases on the CT scan after completion of chemotherapy.

SUMMARY:
The currently developed implementation study aims to evaluate if a patient-led home-based follow-up approach is successful, improves quality of life, reduces anxiety and lessens fear of cancer recurrence during the years after treatment of certain types of testicular cancer.

DETAILED DESCRIPTION:
Testicular cancer represents 1% of male neoplasms and 5% of all urological tumours. In 2021, 828 new patients in the Netherlands were diagnosed with testicular cancer. It is the most commonly diagnosed cancer among young men aged 20-39 years in the Netherlands and incidence is rising. Follow-up after treatment of testicular cancer consists of tumour marker assessment during hospital visits and multiple types of imaging at certain time points. Frequent hospital visits have significant impact on patients' lives, as in-hospital visits evoke distress around the time of visits. Home-based follow-up could be beneficial in terms of patients' well-being and societal cost-effectiveness. Furthermore, during the COVID-19 pandemic hospital visitations are minimized to decrease the chance of COVID-19 exposure. Home-based blood sampling will allow patients to stay home and avoid crowded areas such as public transport and the hospital.

Efforts to improve the current standard of follow-up in patients with testicular cancer should focus on ameliorating quality of life and cost-effectiveness. It provides an opportunity to support patients emotionally, to evaluate treatment effects and complications, and to inform them on their individual prognosis. This is especially true considering the growing importance of value-based healthcare and patient reported outcomes in medicine. The investigators therefore propose a patient-led home-based follow-up approach. This follow-up strategy primarily consists of tumour marker level monitoring at home and imaging performed in-hospital, but additional counselling/diagnostic testing remains possible if desired by patients. In this way the investigators hope to meet the individual needs of patients during follow-up and to improve quality of life outcomes, while achieving equal or greater societal cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically confirmed testicular cancer without distant metastasis and treated with curative intent less than 3 months ago:

  1. Non-seminomatous germ cell tumours, stage I low risk:
* No lymphadenopathy or metastases on the postoperative scan.
* Three consecutive blood drawings with normal tumour markers.
* Patients undergoing lymph node dissection as a second curative operation after an orchiectomy, can also be included in case that the postoperative scan shows no residual disease or metastases.

  2. Non-seminomatous germ cell tumours, stage I high risk:
* After completion of one cycle of Bleomycin, etoposide and platinum (BEP).
* Biochemical remission at completion of chemotherapy, meaning three consecutive blood drawings with normal tumour markers.
* No lymphadenopathy or metastases on the CT scan after completion of chemotherapy.

  3. Seminomatous or non-seminomatous germ cell tumours (after chemotherapy) with complete remission.
* Biochemical remission at completion of chemotherapy, meaning three consecutive blood drawings with normal tumour markers.
* No lymphadenopathy or metastases on the CT scan after completion of chemotherapy.
* Scheduled or currently undergoing postoperative surveillance according to national and European guidelines.
* Signed informed consent.

Exclusion Criteria:

* Patients with aberrant levels of LDH preoperatively (LDH >248 U/L).
* Patients enrolled in other studies that require strict adherence to any specific follow-up practice with regular imaging - yearly or more frequent - of the abdomen and/or thorax
* Patients with comorbidity or other malignancy that requires imaging of the abdomen and/or thorax every year or more frequent
* Inability to complete the questionnaires due to illiteracy and/or insufficient proficiency of the Dutch language

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are 18 years or older who received curative intent surgical treatment for testicular cancer, and who (will) undergo postoperative surveillance are eligible. Patients can be included up to 3 months after curative treatment.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Successful implementation | Year 8 (after the last follow-up moment of the last included patient)
  Patient-led follow-up will be considered successful if the used optional follow up rate is below 75%.

SECONDARY OUTCOMES:
Successful home-based sampling | Year 8
  Defined as 25% or more of all scheduled or optional tumour marker assessments actually performed in blood collected by the patients themselves using the self-administered blood-sampling kit
Quality of life of testicular cancer patients | Year 8
  Measured by the EORTC Core Quality of Life questionnaire (QLQ-C30). All scales and single-item measures range from 0-100 and are calculated using their respective formulas. Higher scores mean a better outcome.
Health-related quality of life | Year 8
  Measured by the EORTC Quality of Life Questionnaire - Testicular Cancer Module (EORTC QLQ-TC26). All scales and single-item measures range from 0-100 and are calculated using their respective formulas. Higher scores mean a better outcome.
Momentary quality of life | Year 8
  Measured by ecological momentary assessment using the Global health status of the EORTC QLQ-C30. The 2 items are scored on a Likert-scale from 1 to 7. Higher scores mean a better outcome.
Anxiety | Year 8
  Measured by The State-Trait Anxiety Inventory: Six-Item Short-form (STAI-6). The STAI-6 comprises of 6 items, each scored on a Likert-scale from 1-4. The final score ranges from 20-80 and is calculated by adding up the score of all single items (positive items are reverse scored) and multiplying by 20/6. Higher scores mean a better outcome.
Fear of cancer recurrence | Year 8
  Measured by the Assessment of Survivor Concerns - Cancer Worry subscale (ASC-CW). The total score is calculated by adding up the individual items and ranges from 3-12. Higher scores mean a worse outcome.
Cost-effectiveness of a patient-led home-based follow-up | Year 8
  The primary effect measure for the economic evaluation will be quality of life, using the The European Quality of Life Five Dimension Five Level Scale (EQ-5D-5L) as a basis for measuring utility. The EQ-5D-5L consists of five levels (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), each scored on a Likert-scale from 1-5 and a visual analogue scale (VAS) scored from 0-100. The total score can be converted into an index value to be used in QALY analysis by ways of an index value calculator taking into account country-specific reference values.
Relation between coping style and follow-up preferences | Year 8
  Measured by the Threatening Medical Situations Inventory (TMSI). Total monitoring and blunting scores are obtained by summing up the relevant items, ranging from 12-60.
Satisfaction of the patient-led home-based follow-up | Year 8
  By a two-item questionnaire at the last follow-up. The first question about satisfaction consists of a scale from 1 to 10. Higher score means a better outcome. The second question is an open question whether the patient has ideas to improve the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk J. Grünhagen, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No